CLINICAL TRIAL: NCT02000479
Title: Influence of Exercise Therapy on Insulin Resistance in Patients With Heart Failure
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hasselt University (Other)
Collaborators: Jessa Hospital (Other)
Responsible Party: Principal Investigator, Bert Op't Eijnde, prof. dr., Hasselt University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 11.11/cardio11.01
Record Dates: First submitted 2013-11-27; First posted 2013-12-04 (Estimated); Last update posted 2013-12-10 (Estimated); Status verified 2013-12

CONDITIONS: Chronic Heart Failure

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- training (Experimental): 12 weeks (2 x 6 weeks) of combined exercise training programme (supervised)
  Interventions: Other: training
- Control (No Intervention): Continued usual care, habitual lifestyle

INTERVENTIONS:
Other: training
  Other Names: 12 weeks of combined exercise training
  Arms: training

SUMMARY:
The purpose of this study is to investigate the effects of a combined training programme on insulin resistance, exercise tolerance, muscle strength, body composition and cardiac function in chronic heart failure patients.

It is assumed that the above mentioned clinical parameters will improve due to physical exercise.

DETAILED DESCRIPTION:
1. Background and study aims During the last decades, the prevalence of (pre)diabetes but also of chronic heart failure (CHF) has increased dramatically. Somehow, both conditions are linked, but the mechanisms involved have not been completely clarified yet. It is clear that the presence of (pre)diabetes in CHF patients affects morbidity and mortality. Although feasibility, safety and beneficial effects of exercise training in CHF are generally acknowledged, its effects on insulin resistance are not well understood. Therefore, the presented study aims to investigate the effect of ET on insulin resistance and the possible link with cardiac function, exercise tolerance, muscle strength and body composition in CHF patients.
2. What does the study involve?

   A randomized controlled study (n=30) will be performed over a period of 12 weeks. Following study inclusion, baseline measurements will be performed in 1 week. They include:
   * a maximal exercise test on a bicycle ergometer to assess exercise tolerance,
   * two oral glucose tolerance tests to assess fasting and post-exercise insulin resistance,
   * a venous blood sample to determine HbA1c, blood lipids, BNP,
   * a muscle strength measurement on a isokinetic dynamometer,
   * assessment of body composition via dual energy x-ray absorptiometry,
   * cardiac echography,
   * questionnaires to assess health-related quality of life,
   * a questionnaire (IPAQ) and a pedometer (3 days) to assess physical activity. Following baseline measurements, subjects will be randomized to a control group (CON, n=10) and an exercise intervention group (EX, n=20), matching for gender and reduced/preserved ejection fraction and glucose tolerance. Hereafter, CON will receive usual care and will be advised to maintain their normal lifestyle, EX subjects will be enrolled in a 12-week training program. Following 6 (MID) and 12 (POST) weeks of exercise training including progressive training load adaptations, baseline measurements will be repeated in all patients.
3. What are the possible benefits and risks of participating?

   * Benefits: patients receive a free training program with personal and professional supervision. After completing the study, they receive a report with personal results and evaluation of training effects.
   * Risks: the usual risks of exercise tolerance testing and exercise training in a CHF population are limited because training sessions are held in the supervised conditions of the Jessa hospital and because training characteristics are according to guidelines of the European Society of Cardiology. Exposure to x-rays during body composition assessment is very low, almost negligible.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of chronic heart failure for at least 6 months
* clinically stable (not hospitalized) for more than 3 months prior to the onset of the study
* optimal medical therapy.

Exclusion Criteria:

* any contra-indication for exercise therapy,
* glucose lowering medical therapy,
* active lifestyle with regular physical activity.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2011-04; Primary Completion 2011-06 (Actual); Study Completion 2011-10 (Actual)

PRIMARY OUTCOMES:
insulin sensitivity (insulin profile) | change from baseline to 12 weeks
  glucose and insulin concentration measurements in blood during oral glucose tolerance test

SECONDARY OUTCOMES:
Exercise tolerance | change from baseline to 12 weeks
  maximal cardiopulmonary exercise test on a bicycle ergometer
HbA1c, blood lipids, BNP | change from baseline to 12 weeks
Muscle strength | change from baseline to 12 weeks
  maximal strength and strength endurance tested on a isokinetic dynamometer
Body composition | change from baseline to 12 weeks
  dual energy x-ray absorptiometry
cardiac function | change from baseline to 12 weeks
  echocardiography
Health-related quality of life | change from baseline to 12 weeks
  MLHFQ and Eq5d

CONTACTS AND LOCATIONS:
Overall Officials: An Stevens, dra., Study Chair — Hasselt University